CLINICAL TRIAL: NCT00460941
Title: A Double-blind, Placebo-controlled Titration Study to Investigate the Tolerability, Safety and Pharmacodynamic Profile of a GLP-1 Analogue in Patients With Type 2 Diabetes Mellitus Treated With a Stable Dose of Metformin.
Brief Title: A Titration Study of a Glucagon-Like Peptide-1 (GLP-1) Analogue in Patients With Type 2 Diabetes Treated With Metformin.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC20728
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — taspoglutide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): sc weekly
  Interventions: Drug: Placebo
- Taspoglutide 20mg (Experimental): sc weekly
  Interventions: Drug: Taspoglutide 20mg
- Taspoglutide 20mg-30mg (Experimental): sc weekly
  Interventions: Drug: Taspoglutide 20mg-30mg
- Taspoglutide 20mg-40mg (Experimental): sc weekly
  Interventions: Drug: Taspoglutide 20mg-40mg

INTERVENTIONS:
Drug: Placebo — sc weekly
  Arms: Placebo
Drug: Taspoglutide 20mg — sc weekly
  Arms: Taspoglutide 20mg
Drug: Taspoglutide 20mg-30mg — sc weekly
  Arms: Taspoglutide 20mg-30mg
Drug: Taspoglutide 20mg-40mg — sc weekly
  Arms: Taspoglutide 20mg-40mg

SUMMARY:
This 4 arm study will evaluate the tolerability, efficacy and pharmacodynamics of different doses of a GLP-1 analogue in patients with type 2 diabetes who are treated with a stable dose of metformin. Patients will be randomized to receive either subcutaneous placebo, or subcutaneous GLP-1 analogue (at a dose of 20mg, or a starting dose of 20mg escalating to either 30mg or 40mg), weekly. All patients will continue on their existing metformin treatment regimen throughout the study. The anticipated time on study treatment is <3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* male,and post-menopausal or surgically sterilized female, patients, 18-75 years of age;
* type 2 diabetes mellitus, with stable metformin treatment for >=3 months;
* HbA1c >=7.0% and <=9.5% at screening;
* stable weight +/-10% for >=3 months before screening.

Exclusion Criteria:

* type 1 diabetes mellitus;
* clinically significant gastrointestinal disease;
* treatment with any anti-hyperglycemic medication other than metformin monotherapy during last 3 months;
* use of weight-lowering medications in the last 3 months;
* uncontrolled hypertension;
* previous exposure to GLP-1 or GLP-1 analogues.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients withdrawn because of gastrointestinal effects | Week 9

SECONDARY OUTCOMES:
Mean changes in 24h blood glucose Area Under the Curve (AUC), Fasting Plasma Glucose (FPG), fructosamine, Hemoglobin A1c (HbA1c), body weight, Adverse Events (AEs), laboratory parameters. | Week 9

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (10):
  - Harrisburg, Arkansas
  - Hot Springs, Arkansas
  - Jonesboro, Arkansas
  - National City, California
  - Jacksonville, Florida
  - Madisonville, Kentucky
  - Hyattsville, Maryland
  - Winston-Salem, North Carolina
  - Dallas, Texas
  - Richmond, Virginia
- Australia (2):
  - Adelaide
  - Camperdown
- France (5):
  - Besançon
  - Corbeil-Essonnes
  - Narbonne
  - Paris
  - Poitiers
- Germany (3):
  - Berlin
  - München
  - Neuss
- Mexico (4):
  - Chihuahua City
  - Culiacán
  - Monterrey
  - Tampico
- Lima, Peru
- Ponce, Puerto Rico

REFERENCES:
- [Derived] Ratner R, Nauck M, Kapitza C, Asnaghi V, Boldrin M, Balena R. Safety and tolerability of high doses of taspoglutide, a once-weekly human GLP-1 analogue, in diabetic patients treated with metformin: a randomized double-blind placebo-controlled study. Diabet Med. 2010 May;27(5):556-62. doi: 10.1111/j.1464-5491.2010.02990.x. PMID 20536952